CLINICAL TRIAL: NCT02796495
Title: Natural Sensory Feedback for Phantom Limb Modulation and Therapy
Brief Title: Use of Hand Prosthesis With Direct Nerve Stimulation for Treatment of Phantom Limb Pain
Acronym: EPIONE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been completed in terms of duration but no patient has been recruited during this time
Sponsor: Prof. Wassim Raffoul (Other)
Collaborators: Aalborg University Hospital (Other); University of Freiburg (Other); Université Montpellier (Other); Lund University (Other); Indiana University School of Medicine (Other); Novosense AB (Industry); Mxm-Obelia (Industry); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other); Catholic University of the Sacred Heart (Other); Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Prof. Wassim Raffoul, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-602547-7; 602547 (Other Grant/Funding Number: FP7-HEALTH-2013-INNOVATION)
Record Dates: First submitted 2016-05-30; First posted 2016-06-10 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Phantom Limb Pain
Keywords: Neuroplasticity; Sensory Feedback; Nerve stimulation; Robotic Hand
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Operation of hand prosthesis with direct nerve stimulation (Experimental): A system composed by the integration of the following non-CE marked medical devices specifically designed for the study will be used in one or two amputees:
  * STIMEP (multichannel electrical stimulator for the peripheral nervous system; AXONIC)
  * TIME-4H Intraneural Electrodes (ALBERT-LUDWIGS-UNIVERSITAET FREIBURG)
  * Sensorized Hand Prosthetics for amputees IH2 Prosthetic Azurra Prensilia (Prensilia Ltd.)
  * Prosthetics sensorized hand for amputees DLR/HIT Hand II (Wessling Robotics)
  * ODROID software integration within the afferent and efferent bi-directional control of the robotic hand
  * The EPIONE Psychophysical Testing Platform software for stimulator control
  Interventions: Device: Operation of hand prosthesis with direct nerve stimulation

INTERVENTIONS:
Device: Operation of hand prosthesis with direct nerve stimulation — Four TIME-4H electrodes will be implanted in the median and ulnar nerves of the amputees. The electrodes will be connected with the STIMEP electrical multichannel stimulator. The stimulator will be connected with one of the two sensorized hand prosthesis. Afferent and efferent signals will be elaborated and integrated by the ODROID software.
  The amputees will be able to control the prosthetic hand movement and receive a sensory feedback from the prosthesis sensors.
  The use of the prosthesis during different tasks will be considered the intervention.

SUMMARY:
Phantom limb pain (PLP) is a frequent consequence of amputation, and it is notoriously difficult to treat. Amputation usually follows traumatic injuries or surgery following vascular diseases, diabetes, osteomyelitis or tumours in cases where the loss of the limb is required for the survival of the patient. The loss of a limb or other body parts is usually followed by the sensation that the lost body part is still present and can be felt. These phenomena are called, respectively, phantom awareness and phantom sensation. In 50-80% of amputees neuropathic pain develops in the lost limb also referred to as phantom limb pain (PLP). PLP can be related to a certain position or movement of the phantom limb, and might be elicited or worsened by a range of physical factors (e.g. changes in the weather or pressure on the residual limb) and psychological factors (e.g. emotional stress). It is well known that most treatments available for PLP today, such as pharmacological, surgical, anaesthetic, psychological and other, are ineffective.

Today it is believed that phantom limb pain may be related to changes in the cortex of the brain. There is evidence that these changes may be modulated - or even reversed - by providing sensory input to the stump or amputation zone. For example, cortical reorganization and alleviation of phantom limb pain has been observed in amputees following intense use of a hand prosthesis. However, there is no consistent knowledge on which type of peripheral sensory feedback may be effective in affecting the cortical plasticity or on how to best apply the sensory feedback.

The aim of the proposed research is to create natural, meaningful sensations through providing invasive sensory feedback (i.e. electrical stimulation through intraneural implantation of electrodes) and the effectiveness to alleviate phantom limb pain and restore the cortical neuroplastic changes.

DETAILED DESCRIPTION:
In the current study, which will take place at the Lausanne University Hospital (CHUV, Centre Hospitalier Universitaire Vaudois), 1-2 hand amputated patients experiencing severe PLP will be enrolled and implanted with intraneural nerve electrodes in the arm stump for up to maximal 6 months.

Nerve electrodes will be implanted in two nerves of the arm stump. During daily stimulation sessions the electrodes will be connected to an external stimulator via transcutaneous leads. During the sessions, selective nerve stimulation will be performed. The amputee patient will experience this as sensations (movement, touch, temperature, vibration etc.) originating from the phantom limb. While implanted, the investigators will investigate how well they can induce these sensations and they will provide a stimulation therapy, which consist of stimulation activities and therefore requires the patient to focus on the evoked sensations. Prior to, during and following therapy a series of assessments (standardized across all EPIONE partners to enable comparison) will be conducted to relate therapy with PLP, cortical organization, the mental state etc. of the patient.

Timing of clinical assessments is conducting in the following phases:

1. First visit
2. Pre-screening visit
3. Baseline and Entry
4. Implantation
5. Intervention period: intensive therapy, preliminary outcome, semi-intensive therapy, monitoring
6. Outcome
7. Follow-up
8. Explantation

Procedures are standardized across international EPIONE partners (which carry out different interventions, but similar assessments), to enable comparison between treatment modalities.

Phase 1: First visit. The subject is invited to a meeting with the principal investigator and one of the senior researchers involved in the study to be informed about the experiment. Only the PI, who is a medical doctor, will be allowed to answer health and medical related questions.

Phase 2: Pre-screening. This phase is conducted before the start of the experiment but after the subject has signed the informed consent form. Via questionnaires, tests and interviews it is evaluated if the subject fulfills the inclusion criteria in relation to physical health (able to undergo surgery), depression, normal range of IQ and PLP. The principal investigator will evaluate the results and decide whether the subject should be included or excluded.

Phase 3: Baseline and Entry. This phase aims to determine the stability and intra-subject variability of the pain sensations without treatment. The measure control for the daily variability in pain, assessment scoring variability, site-to-site variability and inter subject variability in the "before intervention" state. These variances will be used in the analysis to estimate baseline noise in the measure. In addition to the questionnaires used for quantifying the perceived phantom limb pain and sensation, the last week before implantation includes the application of cortical mapping methods (EEG and fMRI). During all phases of the study the subject is required to fill out a diary before going to bed about the development of PLP during the day.

Phase 4: Implantation. After the initial phases the patient is implanted with 4 TIME-4H (Transverse Intrafascicular Multichannel Electrode Version 4 for Human) electrodes. Surgical implantation of the TIME-4H electrodes is conducted under full anaesthesia. During the operation, the median and the ulnar nerves are freed through an incision of 20 cm on the medial aspect of the upper-arm. The fascicles of both nerves are dissected free for a couple of centimetres at the level where the TIME-4H electrodes are to be implanted. Four TIME-4H electrodes are pulled into the fascicles of the nerves using the attached needle and thread, two TIME-4H in each nerve. The electrodes are anchored to the nerve using the dedicated anchoring points of the TIME-4H. After placing the electrodes the electrical integrity of each TIME-4H electrode is tested, before closing the wound. Wires are lead out through the skin and the wound is closed. During surgery the subject is treated with prophylactic antibiotics. Prophylactic antibiotics are not administered later in the study due to the risk of the development of resistance. After the implantation the subject is offered to stay at hospital to enable routine assessment of the surgical outcome as long as the PI judges it necessary. The subject will routinely have the wound where the wires exit the arm cleaned and treated to reduce the risk of infection. This will be conducted by a nurse who is member of the project group. The subject will receive training in treating/cleaning the wound and also in what symptoms to be aware of.

Phase 5: Intervention. One week after the surgery, the patient will start daily sessions of nerve stimulation. Therapy of PLP and sensations are assessed via questionnaires prior to and following the stimulation therapy. Several assessments are conducted during this phase with the purpose of characterizing the sensations which can be evoked and to provide sensory stimulation therapy with the aim of alleviating the phantom limb pain. Programs of stimulation will be performed every day (weekends excluded) for up to 3 hours per day according to the daily experimental aims and the compliance of the patient.

The experience will last between 12 and maximum 20 weeks and will be divided in four different phases:

1. Intensive therapy (from 1st to 4th weeks); during this period the experiments will be carried out every day, from Monday to Friday;
2. Preliminary outcome (5th week); during this week, the experiment will be carried out every day, from Monday to Friday; It will consist of questionnaires and cortical mapping (EEG and fMRI).
3. Semi-intensive therapy (from 6th to 11th weeks); during this period the experiments will be carried out only two days per week, Monday and Tuesday (or two other consecutive days of week that the patient would prefer);
4. Monitoring (from 12th week to the end of the experiment, but no later than 20th week); during this period the experiments will be carried out only once a week on Monday (the day could be changed according to the possibilities of the patient and the working team); during this period the weekly evaluation will be performed only if, in case of success of the trial in treating the PLP, the VAS score will became 2 points greater than the minimum score achieved during the previous periods of the trial, or if other types of necessities connected to implant use would occur.

   A cortical mapping (EEG and fMRI) is scheduled to be carried out during the preliminary outcome and at the end of the therapy (during phase 6).

   Stimulation is performed with the aim of inducing meaningful sensory input to the subject and thereby inducing a normalization of the cortical organization and alleviation of PLP. This is sought accomplished by performing activities (program) which reintroduce the missing limb into the subject's body image.

   The program 1 (Pr1) of the experiment will be performed in order to characterize each channel of the TIME-4H electrodes. The Pr1 will be performed:
   * during the intensive phase: • the first three days of the first week after the implant; • the first day in the following weeks (in order to record possible changes of the location, type and strength of the generated sensation and of the lower threshold and upper limits of the charge, over the weeks);
   * during the semi-intensive phase: • the first day of the weeks (in order to record possible changes of the location, type and strength of the generated sensation and of the lower threshold and upper limits of the charge, over the weeks);
   * during the monitoring phase: • the day of the week when the experiment will be carried out (in order to record possible changes of the location, type and strength of the generated sensation and of the lower threshold and upper limits of the charge, over the weeks). Only if there is observed change in the stabilized map, and only over the active sites where the change is observed the mapping will be re-executed.

   The program 2 (Pr2) of the experiment will be aimed at measuring the impedance of the patient and electrode system with the purpose of characterizing it, to investigate possible changes in consecutive days and to eventually correlate it to changes of the lower threshold and upper limits of current during the same period. The Pr2 will be performed:
   * during the intensive phase:

     • the first day of each week
   * during the semi-intensive phase:

     • the first day of the weeks
   * during the monitoring phase: • the day of the weeks when the experiment will be carried out

   The program 3 (Pr3) will be aimed to explore different strategies of simultaneous asynchronous or synchronous multichannel electrical intraneural stimulation. This program will be performed with the aim of trying different combinations of channels and to identify the best pattern to treat the phantom limb pain of the enrolled patients. The Pr3 will be performed:
   * during the intensive phase:

     • the last two days of the first week after the implant;

     • the second day of the following weeks
   * during the semi-intensive phase: • the first day of the weeks
   * during the monitoring phase: • the day of the weeks when the experiment will be carried out. During the treatment program (Tr), the investigators will test the possibility to drive the stimulation produced by electrical stimulator with the transformed signals from sensors in (or over) the robotic hand, which is voluntarily controlled by the user.

   More specifically, the investigators will ask the patient to perform several tasks (depending on capacity, availability and motivation):
   1. Execution of different force levels (up to 8 levels) with the hand prosthesis
   2. Identification of objects physical properties
   3. Embodiment tests
   4. Functional improvement tests

   The Tr will be performed:

   - during the intensive phase:
   * from the third to the fifth day of the second week;
   * every day of the following weeks - during the semi-intensive phase:
   * both days of the trial - during the monitoring phase:
   * the day of the week when the experiment will be carried out

   Phase 6: Outcome. After the therapy a series of assessments (questionnaires and cortical mapping) are performed to evaluate the effect of therapy. No stimulation therapy is conducted during the outcome and the following follow-up phase.

   Phase 7: Follow-up. During the follow-up phase it will be assessed how long time it takes for any effects of pain alleviating to wear off (questionnaires).

   Phase 8: Explantation. In the event of infection, blushing, swelling, pain or other complications which render continuous implantation impossible, the electrodes will be explanted and the subject treated with antibiotics. Explantation of the TIME-4H electrodes may be conducted at the end of the therapy phase. Explantation will be carried out under full anaesthesia. Access is obtained via an insertion made through the skin on the medial side of the upper arm. The TIME-4H electrodes are dissected free, thread cut and the implant pulled out of the nerve and removed. Following the explantation normal wound treatment will be conducted and the stitches removed according to standard procedures.

   The study duration for a subject will be limited by the maximum TIME-4H implantation duration, which has been set to 6 months maximum.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transradial amputation.
* Amputation should be in the chronic, stable phase, such that the stump has healed and the person apart from eventual phantom pain (PLP) is healthy and able to carry out experiments.
* Other treatments for PLP tried with poor results.
* Patient accepts the study protocol as explained by the physician.
* The subject experienced intractable PLP of more than 6 on NRS or VAS (0-10 scale). The frequency of PLP episodes presents more than once a week.

Exclusion Criteria:

* Cognitive impairment
* Current or prior psychological impairments: Major personality disturbance (i.e. borderline, antisocial), Major depression, Bipolar I.
* Pregnancy
* History of or active substance abuse disorder
* Acquired brain injury with residual impairment
* Intellectual Disability (IQ < 70)
* Prior neurological or musculoskeletal disease
* Current or prior dermatological conditions
* Excessive sensitivity to electrical stimulation with surface electrodes. People afraid of electrical stimulation or pain.
* People with other diseases which may affect the function of the nervous system. (Diabetes, HIV, Renal Failure)
* Patients implanted with pacemakers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain (questionnaires) | Change in phantom limb pain perception during the all study (from baseline to maximum 6 months)
  The pain intensity will be assessed using visual analog scale (VAS)
Cortical reorganization (fMRI) | Change in cortical reorganization before and at the end of treatment (from baseline to maximum 6 months)
  The cortical response to peripheral stimulation will be tracked using fMRI

SECONDARY OUTCOMES:
Phantom limb pain (questionnaires) | Change in neuropathic pain symptoms during the all study (from baseline to maximum 6 months)
  The pain symptoms will be assessed using the Neuropathic Pain Symptom Inventory (NPSI)
Cortical reorganization (EEG) | Change in cortical reorganization before and at the end of treatment (from baseline to maximum 6 months)
  The cortical response to peripheral stimulation will be tracked using EEG

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Raffoul, Professor, Principal Investigator — University Hospital Lausanne CHUV
Locations (1):
- University of Lausanne Hospital CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The laws on protection and data sharing is currently being analysed by one of the consortium partners